CLINICAL TRIAL: NCT05599763
Title: Real-life Study Evaluating the Performance of 2% Aqueous Eosin in Children With Diaper Rash
Brief Title: Multicenter, National, Observational, Prospective, Real-life Study Evaluating the Performance of 2% Aqueous Eosin in Children With Diaper Rash
Acronym: EA2
Status: Completed | Type: Observational
Sponsor: Cooperation Pharmaceutique Francaise (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A01221-42
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Diaper Rash
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being conducted to provide updated clinical data on safety and performance (demonstrated previously for CE marking under the Medical Devices Directive) Cooper Aqueous Eosin 2%. This is an observational study conducted under real-life conditions and as part of post-marketing surveillance activity for a device that has been on the market for a long time and a well-established technology, in accordance with the Medical Devices Regulations 2017 /745 (MDR) and MDCG 2020-6 guidelines.

The study will be a multicenter, national, observational, prospective study, with a 7-day follow-up (+/- 2 day). 60 patients are scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Children under 24 months
* With diaper rash for which a prescription for 2% aqueous eosin in a 50 ml vial is made
* SSDDS score >= 3/6
* Not requiring hospitalization
* Written consent of one of the parents
* Affiliated with social security
* Acceptance of one of the parents to participate in a visit on day 7 in the office or, in case of impossibility, with video/internet consultation or with consultation by phone and sending a photo in this case by the parent(s).

Exclusion Criteria:

* Antibiotic therapy in progress or prescribed on day 0, or other local therapeutic topicals prescribed on day 0
* Children with wounds or likely to be allergic to 2% aqueous eosin or to one of the components of 2% aqueous eosin.
* Ongoing diarrhoea (change in the consistency of stools (loose or watery) and / or an increase in the number (≥ 3 stools / day).

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients seen in consultation by French general practitioners and pediatricians
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with an SSDDS score < 3/6 or an improvement of at least 2 points | at day 7 +-2 days
  The SSDDS (Scoring System for Diaper Dermatitis Scale) score is a severity score : the sum of the scores for four areas: severity of erythema and irritation (score from 0 to 3), extension (0 to 1), presence of papules or pustules (0 to 1) and open skin (0 to 1). The possible scores range from 0 (fair skin) to 6 (extensive diaper rash including intense erythema, papules or pustules and open skin with lesion of the dermis).

SECONDARY OUTCOMES:
Percentage of patients completely cured | at day 7 +/-2 days
Healing time according to parent | up to 9 days
Change of the SSDDS score between day 0 and day 7 | at day 7 +/-2 days
  The SSDDS (Scoring System for Diaper Dermatitis Scale) score is a severity score : the sum of the scores for four areas: severity of erythema and irritation (score from 0 to 3), extension (0 to 1), presence of papules or pustules (0 to 1) and open skin (0 to 1). The possible scores range from 0 (fair skin) to 6 (extensive diaper rash including intense erythema, papules or pustules and open skin with lesion of the dermis).
Change in associated signs between day 0 and day 7 | at day 7 +/-2 days
Assessment of tolerance | at day 7 +/-2 days
  Tolerance is measured by adverse events reported
Assessment of compliance | at day 7 +/-2 days
  According to the judgment of the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric HUET, Principal Investigator — CHU DIJON
Locations (1):
- Multiple locations, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: No